CLINICAL TRIAL: NCT02962843
Title: Evaluation of the Incredible Years Teacher Classroom Management Program in Norwegian School and Day-care Settings: Changes in Students' (6-8 Year) and Children's Behavior (3-6 Year)
Brief Title: Evaluation of the IY TCM Program in Norwegian School and Day-care Settings
Acronym: IYTCMNOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UTromso 2009/655 (REK)
Record Dates: First submitted 2016-10-28; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Behavior Problem
Keywords: Behavior Problem; Social Competence; Student; Children
MeSH Terms: conditions — Mental Disorders; Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IY TCM (Experimental): Incredible Year (IY) Teacher Classroom Management (TCM) training, 6 full-day workshops (42 hours)
  Interventions: Behavioral: IY TCM
- Comparison (No Intervention): No Incredible Year (IY) Teacher Classroom Management (TCM) training.

INTERVENTIONS:
Behavioral: IY TCM — The Incredible Years Teacher Classroom Management program is a manualized program for teachers and staff in school and day-care settings to strengthen teacher classroom management strategies, to reduce negative behavior and promote prosocial behavior, as well as school readiness in children. Two qualified IY TCM group-leaders (facilitators) train teachers and staff in groups through six full-day workshops (a total of 42 hours).Workshop 1: Building Positive Relationships with Students, Workshop 1b: Preventing Behavior Problems -The Proactive Teacher, Workshop 2: The Importance of Teacher Attention, Coaching and Praise, Workshop 3: Motivating Children Through Incentives, Workshop 4 & 5: Decreasing Inappropriate Behavior and Workshop 6: Emotional Regulation, Social Skills & Problem Solving.
  Arms: IY TCM

SUMMARY:
The purpose of this study is to evaluate whether training teacher and staff in the Incredible Years (IY) Teacher Classroom Management (TCM) program reduce behavior problems and promote social competence in student aged 6-8 years (school) and in children aged 3-6 year (day-care). To examine group differences from baseline to 8-9 months after, a quasi-experimental control group design with pre- and post-measurements was used.

DETAILED DESCRIPTION:
Evaluation of the Incredible Years (IY) Teacher Classroom Management (TCM) program implemented as a school-wide preventive intervention in regular school and day-care settings, have the potential to change negative behaviors in children aged 3 - 8 year. Forty-four schools were recruited; comprising 1518 students aged 6-8 year, and 91 day-care units comprising 1049 children aged 3-6 year. Multilevel analyzes were used to examine group differences pre-post changes for behavior problems measured with the Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R) and the Teacher Report Form (TRF), as well as group differences pre-post change for social behavior measured the Social Skills Rating System (SSRS). For secondary findings, group differences pre-post changes for teacher- student and teacher-children relationship were measured with the Student-Teacher Relationship Scale (STRS) (teachers N= 444), and teacher-parents interactions were measured with the Teacher-Parent Involvement Questionnaire (INVOLVE-T/P) (parents N = 2109), as well as group differences pre-post change for teachers self- and collective efficacy measured the Norwegian Teacher Self-Efficacy Scale (NTSES) and the Collective Efficacy Scale (CES) (teachers N = 3240).

ELIGIBILITY:
Inclusion Criteria:

* Schools who met predefined criteria for program implementation of IY TCM (intervention) and school who not have implemented any IY program (comparison).
* Students/children aged 3-8 year (until 7 randomly selected from each class) with parents who speak Norwegian.
* Teachers and staff who worked with students/children aged 3-8 years.

Exclusion Criteria:

* Schools who did not met predefined criteria for program implementation of IY TCM.
* Students/children aged 3-8 year with parents who did not speak Norwegian.
* Teachers and staff who did not worked with students/children aged 3-8 years, and who have known the students/children for fewer than 3 weeks.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5807 (Actual)
Dates: Start 2009-08; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in behavior for student 6-8 year measured with the Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R). | From baseline to 8-9 months after.
  The Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R) is a 38-item scale where teacher rate the current frequency and severity of various behavior in student, and whether or not the behavior is currently a problem.
Change in behavior for student 6-8 year measured with the Teacher Report Form (TRF). | From baseline to 8-9 months after.
  The Teacher Report Form (TRF) consist of 118 item and where teacher rate the degree of emotional and behavioral problems observed in students aged 6-18, and the student academic performance and adaptive function. The Total problem scale forms the basis for various subscales for syndromes or clusters of problems areas.
Change in behavior for student 6-8 year measured with the Social Skills Rating System (SSRS). | From baseline to 8-9 months after.
  The Social Skills Rating System (SSRS) contains of 30 items and where teacher rate how often the student show specific social skills, as well as how important the teacher finds these skills for his/her work in classroom or for the student's success in classroom.
Change in behavior for student 6-8 year with severe behavior problems measured with the Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R). | From baseline to 8-9 months after.
  The Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R) is a 38-item scale where teacher rate the current frequency and severity of various behavior in student, and whether or not the behavior is currently a problem.
Change in behavior for student 6-8 year with severe behavior problems measured with the Teacher Report Form (TRF). | From baseline to 8-9 months after.
  The Teacher Report Form (TRF) consist of 118 item and where teacher rate the degree of emotional and behavioral problems observed in students aged 6-18, and the student academic performance and adaptive function. The Total problem scale forms the basis for various subscales for syndromes or clusters of problems areas.
Change in behavior for student 6-8 year with severe behavior problems measured with the Social Skills Rating System (SSRS). | From baseline to 8-9 months after.
  The Social Skills Rating System (SSRS) contains of 30 items and where teacher rate how often the student show specific social skills, as well as how important the teacher finds these skills for his/her work in classroom or for the student's success in classroom.
Change in behavior for student 6-8 year with severe behavior problems measured with the Student-Teacher Relationship Scale (STRS). | From baseline to 8-9 months after.
  The Student-Teacher Relationship Scale (STRS) consists of a 15-item scale and assess teacher perceptions of two features of their relationships with their students: closeness and conflict.
Change in behavior for children 3-6 year without and with severe behavior problems measured with the Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R). | From baseline to 8-9 months after.
  The Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R) is a 38-item scale where teacher rate the current frequency and severity of various behavior in student, and whether or not the behavior is currently a problem.
Change in behavior for children 3-6 year without and with severe behavior problems measured the Caregiver-Teacher Report Form (CTRF) | From baseline to 8-9 months after.
  The Caregiver-Teacher Report Form (CTRF) rated by teachers for children aged 1½-5, and obtain teachers ratings of 99 problem items plus descriptions of problems, disabilities, what concerns respondents most about the child, and the best things about the child.
Change in behavior for children 3-6 year without and with severe behavior problems measured the Social Competence and Behavior Evaluation Scale (SCBE) . | From baseline to 8-9 months after.
  The Social Competence and Behavior Evaluation Scale (SCBE) is a 30-item questionnaire where teacher rate children behavioral problems (externalizing and internalizing) and social competence.

SECONDARY OUTCOMES:
Change in teacher-student relationship for student 6-8 year measured with the Student-Teacher Relationship Scale (STRS). | From baseline to 8-9 months after.
  The Student-Teacher Relationship Scale (STRS) consists of a 15-item scale and assess teacher perceptions of two features of their relationships with their students: closeness and conflict.
Change in teacher-parents interactions for student 6-8 year measured with the Teacher-Parent Involvement Questionnaire (INVOLVE-T). | From baseline to 8 - 9 months after.
  Teacher-Parent Involvement Questionnaire (INVOLVE-T) consist of 20 items and addresses the degree of parental involvement in school based on teacher ratings.
Change in teacher self-efficacy measured with the Teacher Self-Efficacy Scale (student 6-8 year). | From baseline to 8 - 9 months after.
  The Teacher Self-Efficacy Scale refers to the individual teacher ideas of their own ability to accomplish the tasks they are given as a teacher. It is a 24 item scale and consisting of six subscales. The six subscales are instruction, adapting education to individual student's needs, motivating students, keeping discipline, cooperating with colleagues and parents, and coping with changes and challenges.
Change in collective teacher efficacy measured with the Collective Teacher Efficacy Scale (student 6-8 year). | From baseline to 8 - 9 months after.
  The Collective Teacher Efficacy Scale refers to the teacher beliefs about the collective capability of the organization to influence student achievement. Measures the perceived collective teacher efficacy (7 items), external control scale (5 items) and strain factors (4 items).
Change in teacher self-efficacy and collective teacher efficacy measured with Teacher Observed Problem Behavior in School Environment & Classroom (student 6-8 year). | From baseline to 8 - 9 months after.
  The Teacher Observed Problem Behavior in School Environment & Classroom consists of a 23-item scale measuring teacher responses to problem behavior. This scale consists of five sub factors (positive and supportive responses, responses affected by problem solving and negotiation, moderate behavioral rectifying responses, negative consequences, and formal sanctions) giving two categories of classroom management styles; informal and formal.
Change in problem behavior for students 6-8 year measured with the Behavior in School Environment & Classroom (CES). | From baseline to 8 - 9 months after.
  Behavior in School Environment & Classroom (CES) measures the prevalence of problem behaviour in classroom environment with 20 items, and school environment with 15 items.
Change in teacher self-efficacy and collective teacher efficacy measured with Classroom Climate Scale (student 6-8 year). | From baseline to 8 - 9 months after.
  The Classroom Climate Scale (CCS) is a 14-item scale measuring the quality of the learning environment.
Change in student behavior; generalization effects to home environment for student 6-8 year measured with the Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R). | From baseline to 8 - 9 months after.
  The Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R) is a 38-item scale where teacher rate the current frequency and severity of various behavior in student, and whether or not the behavior is currently a problem.
Change in student behavior; generalization effects to home environment for student 6-8 year measured with the Eyberg Child Behavior Inventory (ECBI). | From baseline to 8 - 9 months after.
  Eyberg Child Behavior Inventory (ECBI) consist of 36 problem behaviors commonly reported by parents of children with conduct problems. The inventory assesses behavior on two dimensions, the frequency of the behavior, and whether or not, the behavior is currently a problem.
Change in teacher-children relationship for children 3-6 year measured with the Student-Teacher Relationship Scale (STRS). | From baseline to 8 - 9 months after.
  The Student-Teacher Relationship Scale (STRS) consists of a 15-item scale and assess teacher perceptions of two features of their relationships with their students: closeness and conflict.
Change in teacher-parents interactions for children 3-6 year measured with the Teacher-Parent Involvement Questionnaire (INVOLVE-T). | From baseline to 8 - 9 months after.
  Teacher-Parent Involvement Questionnaire (INVOLVE-T) consist of 20 items and addresses the degree of parental involvement in school based on teacher ratings.
Change in teacher self-efficacy measured with the Teacher Self-Efficacy Scale (student 3-6 year). | From baseline to 8 - 9 months after.
  The Teacher Self-Efficacy Scale refers to the individual teacher ideas of their own ability to accomplish the tasks they are given as a teacher. It is a 24 item scale and consisting of six subscales. The six subscales are instruction, adapting education to individual student's needs, motivating students, keeping discipline, cooperating with colleagues and parents, and coping with changes and challenges.
Change in collective teacher efficacy measured with the Collective Teacher Efficacy Scale (student 3-6 year). | From baseline to 8 - 9 months after.
  The Collective Teacher Efficacy Scale refers to the teacher beliefs about the collective capability of the organization to influence student achievement. Measures the perceived collective teacher efficacy (7 items), external control scale (5 items) and strain factors (4 items).
Change in teacher self-efficacy and collective teacher efficacy measured with The Teacher Observed Problem Behavior in School Environment & Classroom (student 3-6 year). | From baseline to 8 - 9 months after.
  The Teacher Observed Problem Behavior in School Environment & Classroom consists of a 23-item scale measuring teacher responses to problem behavior. This scale consists of five sub factors (positive and supportive responses, responses affected by problem solving and negotiation, moderate behavioral rectifying responses, negative consequences, and formal sanctions) giving two categories of classroom management styles; informal and formal.
Change in children behavior; generalization effects to home environment for children 3-6 year measured with the Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R). | From baseline to 8 - 9 months after.
  The Sutter-Eyberg Student Behavior Inventory-Revised (SESBI-R) is a 38-item scale where teacher rate the current frequency and severity of various behavior in student, and whether or not the behavior is currently a problem.
Change in children behavior; generalization effects to home environment for children 3-6 year measured with the Eyberg Child Behavior Inventory (ECBI). | From baseline to 8 - 9 months after.
  Eyberg Child Behavior Inventory (ECBI) consist of 36 problem behaviors commonly reported by parents of children with conduct problems. The inventory assesses behavior on two dimensions, the frequency of the behavior, and whether or not, the behavior is currently a problem.

IPD SHARING:
Plan to Share IPD: Undecided
The data for the current study is protected by Norwegian law and cannot be made publicly available at the present moment. The UiT -Arctic University of Norway is in the process of making the metadata available for sharing through the Eutro program.

REFERENCES:
- See also: Related Info — http://dua.uit.no/